CLINICAL TRIAL: NCT06349447
Title: The Therapeutic and Preventive Effects of Light-emitting Diodes (LEDs) Irradiation for Post-inflammatory Erythema and Hyperpigmentation: a Self-controlled
Brief Title: Pilot Study of LED for PIE and PIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanjun Dan (Other)
Responsible Party: Sponsor-Investigator, Yanjun Dan, Department of Dermatology, Huashan Hospital, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-771
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hyperpigmentation
Keywords: photobiomodulation, PIE, PIH, LED
MeSH Terms: conditions — Hyperpigmentation; Mediastinal Emphysema

STUDY DESIGN:
Intervention Model Description: 308 nm LED light was utilized to induce an vivo PIE/PIH model on the thigh of subjects. The irradiation dose was 1.5 MED. Five circular experimental lesions measuring 1.5 × 1.5 cm were selected on the thighs, categorizing into five groups: control group, 830 nm LED treatment group, 590 nm LED treatment group, 830 nm LED prevention group and 590 nm LED prevention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: LED irradiation (Experimental): For therapeutic irradiation, the PIH model was induced on D1, and 830 nm (60 J/cm2, 50 mW/cm2) and 590 nm LED (20 J/cm2, 20 mW/cm2) were irradiated on D0, D1, D3, D6 and D8, respectively. For preventive irradiation, 830 nm and 590 nm LED were irradiated on D0, D1, D3, D6 and D8, respectively, and the PIE/PIH model was induced on D9.
  Interventions: Device: LED
- Control (Active Comparator): the PIH model was induced on D1 and without any LED exposition.
  Interventions: Other: without any LED exposition

INTERVENTIONS:
Device: LED — 308 nm LED light was utilized to induce an vivo PIE/PIH model on the thigh of subjects. The irradiation dose was 1.5 MED. Five circular experimental lesions measuring 1.5 × 1.5 cm were selected on the thighs, categorizing into five groups: control group, 830 nm LED treatment group, 590 nm LED treatment group, 830 nm LED prevention group and 590 nm LED prevention group. 830 nm LED and 590 nm LED were irradiated, respectively. For therapeutic irradiation, the PIH model was induced on D1, and 830 nm (60 J/cm2, 50 mW/cm2) and 590 nm LED (20 J/cm2, 20 mW/cm2) were irradiated on D0, D1, D3, D6 and D8, respectively. For preventive irradiation, 830 nm and 590 nm LED were irradiated on D0, D1, D3, D6 and D8, respectively, and the PIE/PIH model was induced on D9.
  Arms: Experimental: LED irradiation
Other: without any LED exposition — without any LED exposition
  Arms: Control

SUMMARY:
The aim of this study is to explore the effect of medical LEDs (830 nm and 590 nm) in the prevention and treatment of PIE and PIH.

DETAILED DESCRIPTION:
Evidence regarding the efficacy of LEDs for post-inflammatory erythema (PIE) and post-inflammatory hyperpigmentation (PIH) is limited.

The aim of this study was to evaluate the efficacy of 830 nm and 590 nm LED phototherapies on PIE and PIH.

Design of the study:

308 nm LED light (1.5 MED) induced an in vivo PIE/PIH model on the thigh of ten healthy subjects. 830 nm (60 J/cm2) and 590 nm LED (20 J/cm2) were irradiated respectively. For therapeutic irradiation, PIE/PIH model was induced on D1, and LEDs were irradiated on D0, 1, 3, 6 and 8. For preventive irradiation, LEDs were irradiated on D0, 1, 3, 6 and 8 and PIE/PIH model was induced on D9. Erythema index (EI), melanin index (MI), transdermal water loss (TEWL) and C-Cube photography were measured during 10-day follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Asians;
2. 20-65 years old;
3. Fitzpatrick classification III-IV;
4. Sign the informed consent form.

Exclusion Criteria:

1. Have abnormal skin manifestations, such as pigment diseases, photosensitivity diseases and other allergic diseases;
2. Those with a history of abnormal systemic diseases, such as heart disease, liver disease, kidney disease, tumors, and mental illness;
3. Women who are preparing for pregnancy, pregnant or breastfeeding;
4. Have used photosensitizing drugs within two weeks before inclusion in this study;
5. Topical or systemic drugs may be used during this study;
6. bad habits, such as smoking, drinking, etc.;
7. Volunteers who have recently participated in other clinical trials;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
melanin index | at day 8
  The effect of LED treatment on PIH will be estimated by measure by C-CUBE.
erythema index | at day 8
  The effect of LED treatment on PIE will be estimated by measure by C-CUBE.

SECONDARY OUTCOMES:
transepidermal water loss (TEWL) | at day 8
  The effect of LED treatment on skin water loss will be estimated by measure by delfin.
elasticity | at day 8
  The effect of LED treatment on skin elasticity will be estimated by measure by delfin.

CONTACTS AND LOCATIONS:
Overall Officials: Leihong Xiang, professor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No